CLINICAL TRIAL: NCT06991205
Title: Feasibility RCT of Web-based Mind-body Treatment to Enhance Resilience Among Patients With Painful Nontraumatic Upper-extremity Conditions and Commorbid Risky Substance Use
Brief Title: Web-based Mind-body Program to Improve Resilience Among Risky Substance Users With Persistent Upper Extremity Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jafar Bakhshaie (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Jafar Bakhshaie, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P001335; 5K23AT012364-03 (NIH)
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Orthopedic Disorder; Nontraumatic Injury; Upper Extremity Pain; Risky Substance Use
Keywords: Upper Extremity Problem; Risky substance use; Randomized Controlled Trial (RCT); Mindfulness; Nontraumatic conditions; Chronic pain; Psychiatry; Feasibility
MeSH Terms: conditions — Musculoskeletal Diseases; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-TIRELESS (Experimental): A 4-session, asynchronous, web-based mind-body pain and substance use management intervention.
  Interventions: Behavioral: Web-TIRELESS
- Web-MEUC (Active Comparator): Open access to a web-based pamphlet containing brief, educational information and coping techniques.
  Interventions: Other: Web-MEUC

INTERVENTIONS:
Behavioral: Web-TIRELESS — This is a self-administered web-based intervention that consists of 4 on-demand sessions, each ~30 minutes long, that teach mind-body skills, cognitive-behavioral strategies (e.g., reframing, pain and substance use urge surfing), activity pacing, acceptance and commitment skills, and psychoeducation on the association between substance use and pain. The program aims to increase patients' physical and emotional functioning and decrease pain intensity and maladaptive substance use behaviors.
  Arms: Web-TIRELESS
Other: Web-MEUC — An educational information web-based pamphlet, containing brief, summarized information tailored for the respective patient population that follows topics including the trajectory of pain and adaptation after non-traumatic painful upper extremity conditions, the role of relaxation strategies to manage pain, and the importance of returning to engagement in activities of daily living.
  Arms: Web-MEUC

SUMMARY:
The investigator aims to conduct a feasibility randomized controlled trial (RCT) (N=50) to test the feasibility, acceptability, and credibility of an asynchronous web-based mind-body intervention (Toolkit for Resilient Life beyond Pain and Substance Use; Web-TIRELESS) versus web-based minimally enhanced usual care (Web-MEUC) among adult patients with a painful non-traumatic upper-extremity condition(s) (PNUC) and commorbid risky substance use.

Deliverables: [1] Adapt and refine open pilot protocol, patient recruitment, and other study materials. [2] Assess the feasibility, acceptability, and credibility of Web-TIRELESS and Web-MEUC in preparation for future research.

DETAILED DESCRIPTION:
Aim: Conduct a feasibility randomized controlled trial (RCT) (N=50) of Web-TIRELESS versus Minimally Enhanced Usual Care (Web-MEUC)-both of which are web-based-among patients with painful nontraumatic upper extremity conditions and comorbid risky substance use (N=50), to demonstrate the feasibility of recruitment procedures and data collection; and the feasibility, credibility, and acceptability (adherence, retention, fidelity, and satisfaction) of Web-TIRELESS and Web-MEUC. We will use this mixed-methods information to assess the primary outcomes and optimize both programs and study methodology in preparation for research.

Participants are randomized to either Web-TIRELESS or Web-MEUC and given access to the respective program for approximately 5 weeks to review and complete the assigned material. Both groups are given education material to help improve pain and substance use urge coping. There are 3 assessment points consisting of self-report surveys: baseline, post-program, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient adults seeking care in the Hand and Arm Center
2. Diagnosed with a non-traumatic painful upper-extremity condition (NPUC)
3. Pain score > 4 on the Numerical Rating Scale (NRS)
4. Risky substance use (scores >10 and <27 for alcohol, and >3 and <27 for cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opioids, tobacco products, and e-cigarette on The World Health Organization's - Alcohol, Smoking and Substance Involvement Screening Test [WHO-ASSIST])
5. Owns a smartphone, laptop, or computer with internet access
6. Age ≥18yr
7. English fluency
8. Ability and willingness to participate in a live video focus group and the following asynchronous Web-based intervention

Exclusion Criteria:

1. Participation in mind-body or specialized substance abuse treatment in the past 3 months
2. Practice of mindfulness >45 minutes/week in the past 3 months
3. Psychotropic medications (e.g. antidepressants) changed in the past 3 months
4. Serious untreated mental illness (e.g., Schizophrenia)
5. Suicidal ideation with intent or plan
6. Pregnancy
7. Secondary gains that may bias motivation (e.g., pending disability claim),
8. Moderate to severe cognitive impairment (score ≥4 on the Short Portable Mental Status Questionnaire (SPMSQ))
9. History of surgery for the presented NPUC within the past 6 months OR future plans for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Baseline (0 Weeks)
  Assesses the degree to which one believes the intervention will effectively manage their condition, substance use, and related worry. Possible scores range from 3 to 27 for both the credibility and the expectancy subscales. Higher scores represent higher credibility and expectancy.
Client Satisfaction Questionnaire to assess satisfaction with/acceptability of treatment | Post-Test (5 Weeks)
  Participants' satisfaction with treatment received after completion. The score range is 0-12. Higher scores indicate greater satisfaction.
The User Experience Scale to assess participants' satisfaction with (acceptability of) web-based delivery | Post-Test (5 Weeks)
  This measure will assess how well patients like the Wed-based program content and delivery. Total raw scores range from 22 to 110 with higher scores indicating greater satisfaction with the platform.
The percent of patients that agree to participate to assess feasibility of recruitment | Baseline (0 Weeks)
  The percent of eligible patients approached that agree to participate.
Rate at which program was accepted, measured by attendance to assess acceptability of treatment | Post-Test (5 Weeks)
  The proportion of Web-TIRELESS participants who complete > or = 3 of 4 sessions.
Adherence to homework | Throughout intervention completion, an average of 1 month
  Rate of Web-TIRELESS participant's completion of homework assigned throughout the study.
Rate of participant's completion of self-report measures to assess feasibility of assessments | Baseline (0 Weeks), Post-Test (5 Weeks)
  Investigators will report number of patients who complete assessments at each time-point.
Adverse Events | Throughout intervention completion, an average of 1 month
  Any self-reported or observed negative events related to participation.

SECONDARY OUTCOMES:
Graded Chronic Pain Scale (GCPS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  Assesses pain severity and pain-related disability. Total scores range from 0 to 10, with higher scores indicating worse pain severity.
Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  A 30-item measure that assesses disability severity. Scores range from 0 to 100 with higher scores indicating greater disability.
Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depression-Short Form 8a v1.0 | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  An 8-item measure assessing symptoms of depression. Scores range from 8 to 40 with higher scores indicating greater symptom severity
PROMIS Emotional Distress - Anxiety-Short Form 8a v1.0 | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  An 8-item measure assessing symptoms of anxiety. Scores range from 8 to 40, with higher scores indicating greater symptom severity.
Pain Catastrophizing Scale (PCS) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  Assesses magnification, helplessness, and rumination about pain. Scores range from 0 to 52. Higher scores indicate greater pain catastrophizing.
Pain Anxiety Symptoms Scale - Short Form (PASS-20) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  Assesses fear and anxiety related to pain. Scores range from 0 to 100. Higher scores indicate greater pain-related fear and anxiety.
Pain Vigilance and Awareness Questionnaire (PVAQ) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  Assesses preoccupation with or attention to pain. Scores range from 16 to 96. Higher scores indicate greater pain vigilance.
Brief Experiential Avoidance Questionnaire (BEAQ) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  This measure assesses tendencies to avoid unpleasant internal experiences. Scores range from 15 to 90. Higher scores suggest greater avoidance behaviors.
Current Opioid Misuse Measure (COMM) | Baseline (0 Weeks), Post-Test (5 Weeks), Follow-Up (6 Months)
  Assesses risk for aberrant medication-related behavior in persons with chronic pain. Scores range from 0 to 68. Higher scores indicate greater risk for opioid misuse.
The Timeline Follow Back (TLFB) | Throughout intervention completion, an average of 1 month
  Assesses daily estimates of alcohol, cannabis, cigarette, and other drug use during the past week. The range is 0 to 7 days, with higher scores indicating more severe use.
Numerical Rating Scale (NRS) | Eligibility Screening (-1 Weeks)
  Severity of participant's average ans worse pain over the last 3 months using a Likert scale with 0 being no pain and 10 being worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jafar Bakhshaie, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No